CLINICAL TRIAL: NCT00245804
Title: Developmental Dyslexia and Functional Maturation of Auditory Cortex
Acronym: DYS-AUT
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: HOMMET CAROLINE,MD-PHD, INSERM
Other Study IDs: PHRR02/CH/DYS-AUT
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2005-01

CONDITIONS: Developmental Reading Disorder; Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Adult dyslexia: Adult dyslexia
- Minor-Dyslexia: Minor-Dyslexia
- Adult-Control: Adult-Control
- Minor-Control: Minor-Control

SUMMARY:
Developmental dyslexia is a frequent learning disability. The aim of this study is to compare auditory evoked cortical responses to syllables and tones in developmental dyslexia and controls (paired with age, gender). The study is conducted in 3 groups of subjects :8-10 years ; 11-17 years and 18-25 years. We suppose that cortical responses should be different in developmental dyslexia and controls.

ELIGIBILITY:
Inclusion Criteria:

Age (8-10 years ; 11-17 years ; 18-25 years developmental reading disorders (developmental dyslexia) criteria according to Critchley (1970) PIQ > 85 No auditory deficit No psychosis -

Exclusion Criteria:

PIQ < 85 Epilepsy ADHD Stroke, head injury

-

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with developmental reading disorders from 8 to 25 jears. Control groupes with healthy people in de same age
Sampling Method: Probability Sample
Enrollment: 60
Dates: Start 2003-03; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hommet, Principal Investigator — University Hospital of Tours
Locations (1):
- University Hospital of Tours, Tours, France